CLINICAL TRIAL: NCT04591379
Title: Intratumoral Influenza Vaccine for Early Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REG-083-2020
Record Dates: First submitted 2020-09-07; First posted 2020-10-19 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Experimental)
  Interventions: Drug: Influenza Vaccines

INTERVENTIONS:
Drug: Influenza Vaccines — Intratumoral application of an unattenuated influenza vaccine

SUMMARY:
The aim of this explorative phase II clinical trial is to establish the safety and efficacy of intratumoral influenza vaccine in patients with colorectal cancer, as an additive treatment prior to intended curative surgery.

DETAILED DESCRIPTION:
This is an explorative phase 2 clinical trial which will be conducted in two phases. The aim of this study is to establish the safety and efficacy of treating patients with early colorectal cancer with intratumoral influenza vaccine as a down staging and immune response enhancing treatment prior to intended curative surgery.

The first part of the study will be conducted as a pilot study. Six patients with histologically verified or clinically suspicious sigmoid colon cancer who are planned to undergo curative surgery will be included. Patients will be recruited from the Department of Surgery, Zealand University Hospital after their case has been reviewed by the multidisciplinary team (MDT). Standard treatment involves intended curative surgery within two weeks after the diagnosis. The treatment will be performed within a few days and it will be ensured that the experimental treatment will not lead to a significant delay of intended curative surgery.

If the pilot study finishes without violating any stop rules and without any serious adverse events the second part of the study will be initiated. This will be conducted as a phase 2 study where 24 patients with histologically verified or clinically suspicious sigmoid colon cancer and rectal cancer will be included. Patients will be recruited from the Department of Surgery, Zealand University Hospital after their case has been reviewed by the multidisciplinary team (MDT). Standard treatment involves intended curative surgery within two weeks after the diagnosis. The treatment will be performed within a few days and it will be ensured that the experimental treatment will not lead to a significant delay of intended curative surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be mentally capable of understanding the information given.
* Patients must give written informed consent.
* Clinically suspected or histologically verified malignant tumor of the rectum or sigmoid colon.
* Tumor described as passable at index endoscopy.
* Men or women aged at least 18 years.
* Case reviewed by MDT (surgery, radiology, oncology). Case considered curable with standard surgical resection.

Exclusion Criteria:

* Highly inflamed gastrointestinal tissue which is ulcerated and bleeding
* Ongoing immunosuppressive treatment.
* Concurrent treatment with an investigational medicinal product.
* Patients with any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study recruitments.
* Advanced tumor stages, clinical UICC stage IV.
* Indication for neoadjuvant chemoradiation or chemotherapy prior to surgery
* Acute surgical resection.
* Pregnancy
* Any previous allergic reaction to influenza vaccine or constituents, egg and chicken proteins, neomycin, formaldehyde or octoxinol-9
* Acute febrile illness
* Acute infectious disease
* Influenza vaccine administered within 30 days before study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Safety - Adverse reactions are classified according to CTCAE version 4.0 | Day of surgery (day 7-14 after treatment)
  To investigate if intratumoral influenza vaccine is a safe treatment modality for tumor down staging prior to intended curative surgery in patients undergoing treatment for colorectal cancer.
  Adverse events / reactions are recorded from day of treatment (Day 0) until the surgery, as it will be difficult to differ between adverse events/reactions to the experimental treatment or surgery. All adverse events / reactions should be described in medical terminology in the patient's file and recorded in case report forms (CRF). The following information must be recorded: start date/date when observed, severity, any initiated treatment, assessment of the AE if it meets the criteria for SAE, end date, and relationship to study drug. For AEs that meet the criteria for SAE, the outcome must be recorded.

SECONDARY OUTCOMES:
Efficacy - local immunological changes | Pathological specimens from day of treatment (day 0) and surgery (day 7-14 after treatment)
  To investigate if intratumoral influenza vaccine will induce immunologic invasion of the primary tumor This will be analyzed by immunhistochemistry and NanoString

OTHER OUTCOMES:
Efficacy - systemic immunological changes | Blood samples from the day of treatment (day 0), before surgery (day 7-14 after treatment), after surgery (postOP day 1-2) and postoperative follow-up (postOP day 12-16)
  To investigate if the treatment will induce a systemic immunologic response.
Quality of recovery | Assessed before treatment (day 0), before surgery (day 7-14 after treatment), after surgery (postOP day 1) and postoperative follow-up (postOP day 12-16)
  To assess quality of recovery for patients recruited into this trial. A quality of recovery questionnaire (QoR-15) will be given to patients pre- and post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, Professor, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Køge, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Study protocol and informed consent form will be available upon start of recruitment of patients

REFERENCES:
- [Derived] Gogenur M, Balsevicius L, Bulut M, Colak N, Justesen TF, Fiehn AK, Jensen MB, Host-Rasmussen K, Cappelen B, Gaggar S, Tajik A, Zahid JA, Bennedsen ALB, D'Ondes TDB, Raskov H, Saekmose SG, Hansen LB, Salanti A, Brix S, Gogenur I. Neoadjuvant intratumoral influenza vaccine treatment in patients with proficient mismatch repair colorectal cancer leads to increased tumor infiltration of CD8+ T cells and upregulation of PD-L1: a phase 1/2 clinical trial. J Immunother Cancer. 2023 May;11(5):e006774. doi: 10.1136/jitc-2023-006774. PMID 37172969